CLINICAL TRIAL: NCT03551769
Title: A Phase I, Open-label, Fixed-order, Single-dose, 2-Part, Crossover Study to Evaluate the Pharmacokinetics of a Formulation of Tricaprilin (AC-SD-01) Including the Effect of Food on Ketone Body Production in Caucasians and Asians
Brief Title: Pharmacokinetics of Tricaprilin Including Food Effect on Ketone Body Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AC-18-016_FE
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tricaprylin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1, Period 1 (Experimental): Study drug administered concurrently with a standard meal
  Interventions: Drug: tricaprilin; Other: standard meal
- Cohort 1, Period 2 (Experimental): Study drug administered 30 minutes after a standard meal
  Interventions: Drug: tricaprilin; Other: standard meal
- Cohort 1, Period 3 (Experimental): Study drug administered 30 minutes after a high-fat meal
  Interventions: Drug: tricaprilin; Other: high-fat meal
- Cohort 1, Period 4 (Experimental): Study drug administered after an overnight fast
  Interventions: Drug: tricaprilin
- Cohort 2, Period 1 (Experimental): Study drug administered 30 minutes after a standard meal (Asian)
  Interventions: Drug: tricaprilin; Other: standard meal
- Cohort 2, Period 2 (Experimental): Study drug administered after an overnight fast (Asian)
  Interventions: Drug: tricaprilin; Other: overnight fast

INTERVENTIONS:
Drug: tricaprilin — Tricaprilin formulated as AC-SD-01
Other: standard meal — standard meal
  Arms: Cohort 1, Period 1; Cohort 1, Period 2; Cohort 2, Period 1
Other: high-fat meal — high-fat meal
  Arms: Cohort 1, Period 3
Other: overnight fast — fasting for at least 9 hours
  Arms: Cohort 2, Period 2

SUMMARY:
This is a Phase I, single center, open label, fixed-order, crossover, food-effect, pharmacokinetic (PK) study recruiting healthy, adult, male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male, ages 18 - 55
* Able to consume a regular diet and one high fat meal; no specific dietary requirements
* Cohort 2 (Asian subject population) restricted to being of Japanese or Chinese heritage

Exclusion Criteria:

* Presence of any illness or condition that, in the opinion of the investigator might confound the study results or poses risk to the subject
* Has been on a ketogenic diet as supported by review of a food diary
* Has positive Urine Drug Screen or alcohol results at Screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Total ketones | 1 day
  Area Under the Curve (AUC) AUC 0-last
Total ketones | 1 day
  AUC 0 - 4
Total ketones | 1 day
  AUC 0 - 6
Total ketones | 1 day
  AUC 0-8
Total ketones | 1 day
  Maximum Plasma Concentration (Cmax)
B-hydrodxybutyrate | 1 day
  AUC 0-last
B-hydroxybutyrate | 1 day
  AUC 0-4
B-hydroxybutyrate | 1 day
  AUC 0-6
B-hydroxybutyrate | 1 day
  AUC 0-8
B-hydroxybutyrate | 1 day
  Cmax
Acetoacetate | 1 day
  AUC 0-last
Acetoacetate | 1 day
  AUC 0-4
Acetoacetate | 1 day
  AUC 0-6
Acetoacetate | 1 day
  AUC 0-8
Acetoacetate | 1 day
  Cmax

SECONDARY OUTCOMES:
tricaprilin | 1 day
  AUC 0 - last
tricaprilin | 1 day
  AUC 0 - 4
tricaprilin | 1 day
  AUC 0 - 6
tricaprilin | 1 day
  AUC 0 - 8
tricaprilin | 1 day
  Time to maximum concentration (Tmax)
tricaprilin | 1 day
  Cmax
octanoic acid | 1 day
  AUC 0 - last
octanoic acid | 1 day
  AUC 0 - 4
octanoic acid | 1 day
  AUC 0 - 6
octanoic acid | 1 day
  AUC 0 - 8
octanoic acid | 1 day
  Tmax
octanoic acid | 1 day
  Cmax
Computerized Cognitive Battery - Attention | 1 day
  Rapid Visual Information Processing Test
Computerized Cognitive Battery - Episodic Memory | 1 day
  Paired Associates Learning Test
Computerized Cognitive Battery - Working Memory | 1 day
  Spatial Working Memory Test
Computerized Cognitive Battery - Psychomotor Function | 1 day
  Reaction Time Test

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No